CLINICAL TRIAL: NCT02126579
Title: Open Label, Randomized, Phase I/II Study of a Long Peptide Vaccine Plus TLR Agonists for Resected Stage IIb-IV Melanoma. (MEL60)
Brief Title: Phase I/II Trial of a Long Peptide Vaccine (LPV7) Plus TLR Agonists
Acronym: MEL60
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15931; MEL60 (Other: UVA Human Immune Therapy Center)
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Melanoma; Metastatic Melanoma; Mucosal Melanoma
Keywords: melanoma; neoplasms; Poly ICLC; Freund's Adjuvant; Metastatic melanoma; resiquimod; adjuvants; peptide vaccine
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Protein Subunit Vaccines; resiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Arm A (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + IFA administered in one skin location rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: IFA
- Arm B (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC vaccine administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: PolyICLC
- Arm C (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide vaccine administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after the vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: Resiquimod
- Arm D (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: PolyICLC; Other: Resiquimod
- Arm E (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: PolyICLC; Other: IFA
- Arm F (Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + IFA vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: Resiquimod; Other: IFA
- Arm G(Part 1) (Experimental): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC + IFA vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: PolyICLC; Other: Resiquimod; Other: IFA
- Arm E2 (Experimental): Peptide Vaccine (LPV7) + IFA + PolyICLC vaccines administered in one skin location. Each vaccine will be administered in the same skin site for all 6 vaccines.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: Peptide Vaccine (LPV7) + Tetanus peptide; Other: PolyICLC; Other: IFA

INTERVENTIONS:
Biological: Peptide Vaccine (LPV7) + Tetanus peptide — 1.5 mL administered half intradermally and half subcutaneously.
Other: PolyICLC — 1 mL administered half intradermally and half subcutaneously
  Arms: Arm B (Part 1); Arm D (Part 1); Arm E (Part 1); Arm E2; Arm G(Part 1)
Other: Resiquimod — 500 mg applied to vaccine site after vaccine administration
  Arms: Arm C (Part 1); Arm D (Part 1); Arm F (Part 1); Arm G(Part 1)
Other: IFA — 2 mL administered half intradermally and half subcutaneously
  Arms: Arm A (Part 1); Arm E (Part 1); Arm E2; Arm F (Part 1); Arm G(Part 1)

SUMMARY:
The purpose of this study is to learn what effects (good and bad) an experimental vaccine (LPV7) plus tetanus peptide and other substances called polyICLC, resiquimod, and Montanide ISA-51 have on you and your melanoma. We will also look at whether the experimental vaccine and these drugs cause any changes in your immune system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven Stage IIB - IV melanoma rendered clinically free of disease by surgery, other therapy, or spontaneous remission within 6 months prior to registration.

  * Patients may have had melanoma from a cutaneous, mucosal or unknown primary site
  * Patients with small radiologic or clinical findings may be eligible
* Patients with treated brain metastases may be eligible if the following are true:

  * Total number of brain metastases ever is less than or equal to 3
  * The brain metastases have been completely removed by surgery or have been treated completely with stereotactic radiotherapy
  * There has been no evident growth of any brain metastases since treatment
  * No treated brain metastases is greater than 2 cm at the time of protocol entry
* Patients must have at least 1 intact axillary and/or inguinal lymph node basin
* ECOG performance status of 0-1
* Lab parameters as follows:

  * HLA-A1, A2, A3, B35, or B51
  * ANC > 1000/mm3 and Platelets > 100,000/mm3 and Hemoglobin > 9 g/dL
  * AST and ALT up to 2.5 x ULN
  * Bilirubin up to 2.5 x ULN
  * Alkaline Phosphatase up to 2.5 x ULN
  * Creatinine up to 1.5 x ULN
  * HGBA1C level ≤ 7.5%

Exclusion Criteria:

* Patients with melanoma from a uveal or ocular primary site
* Patients currently receiving any systemic therapy within 4 weeks of study registration. Gamma knife or stereotactic radiosurgery must not be administered within 1 week prior to study registration. Patients who are currently receiving nitrosoureas within the preceding 6 weeks.
* Patients who have received CTLA-4, PD-1, PD-L1, CD137, or CD27 within the prior 12 months.
* Patients with known or suspected allergy to any component of the vaccine
* HIV positive or active Hepatitis C virus
* Patients receiving any of the following medications within 4 weeks are excluded:

  * Agents with immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents and topical steroids)
  * Allergy desensitization injections
  * Systemic corticosteroids, administered parenterally or orally. Inhaled steroids (e.g. Advair, Flovent, Azmacort) are not permitted. Topical corticosteroids are acceptable including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex)
  * Any growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
  * Interferon therapy
  * Interleukin-2 or other interleukins
* Other investigational drugs or investigational therapy if currently receiving or have received within 1 month
* Pregnancy or the possibility of becoming pregnant during the study. And women who are breastfeeding.
* Must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. The following are not exclusionary:

  * Presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring NSAID medications
* Patients with a medical contradiction or potential problem with complying with the protocol, in the opinion of the investigator
* Patients with Class III or IV heart disease (according to NYHA classification)
* Patients with a body weight < 110 lbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, Jr., M.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - MDAnderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Patel SP, Petroni GR, Roszik J, Olson WC, Wages NA, Chianese-Bullock KA, Smolkin M, Varhegyi N, Gaughan E, Smith KT, Haden K, Hall EH, Gnjatic S, Hwu P, Slingluff CL. Phase I/II trial of a long peptide vaccine (LPV7) plus toll-like receptor (TLR) agonists with or without incomplete Freund's adjuvant (IFA) for resected high-risk melanoma. J Immunother Cancer. 2021 Aug;9(8):e003220. doi: 10.1136/jitc-2021-003220. PMID 34413169
- See also: NCI website — http://www.cancer.gov/cancertopics/types/melanoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrolling 49 participants across all 7 arms in accord with the study objectives, the study was amended to allow enrollment of an additional cohort on arm E (part 2) as a neoadjuvant vaccine with biopsies pre- and post-vaccine. However, only 1 patient enrolled on part 2 arm E; thus, we closed the study. Analysis of 1 patient would not satisfy the goals of that neoadjuvant component; so, we include data for the part 2 Arm E participant in Arm E for reporting purposes.
Groups:
- Arm A (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + IFA administered in one skin location rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  IFA: 2 mL administered half intradermally and half subcutaneously
- Arm B (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC vaccine administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
- Arm C (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide vaccine administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after the vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  Resiquimod: 500 mg applied to vaccine site after vaccine administration
- Arm D (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  Resiquimod: 500 mg applied to vaccine site after vaccine administration
- Arm E (Part 1 + Part 2): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma (except that the vaccines were administered to the same skin site for the one patient from cohort 2)
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously. (except that the tetanus peptide was not included in the vaccine for the one patient on this arm from cohort 2.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  IFA: 2 mL administered half intradermally and half subcutaneously
- Arm F (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + IFA vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  Resiquimod: 500 mg applied to vaccine site after vaccine administration
  IFA: 2 mL administered half intradermally and half subcutaneously
- Arm G(Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + PolyICLC + IFA vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Resiquimod will be applied to the vaccine site immediately after vaccine administration.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  Resiquimod: 500 mg applied to vaccine site after vaccine administration
  IFA: 2 mL administered half intradermally and half subcutaneously
Period: Overall Study
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1 + Part 2) | Arm F (Part 1) | Arm G(Part 1)
Started | 5 | 7 | 4 | 6 | 16 | 6 | 6
Received at Least 3 Vaccines | 5 | 7 | 4 | 6 | 16 | 6 | 6
Completed (Completed all 6 vaccines) | 5 | 7 | 4 | 5 | 16 | 6 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — disease progression | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm E (Part 1 + 2): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  IFA: 2 mL administered half intradermally and half subcutaneously.
  Except that the last patient, on Part 2 received all 6 vaccines in the same site and did not receive tetanus peptide.
- Total: Total of all reporting groups
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1 + 2) | Arm F (Part 1) | Arm G(Part 1) | Total
Number analyzed (Participants) | 5 | 7 | 4 | 6 | 16 | 6 | 6 | 50
Age, Customized [Median (Full Range); unit: years]
  Median Age | 52 [33 to 62] | 64 [21 to 69] | 64 [44 to 76] | 53 [19 to 67] | 60 [24 to 71] | 56 [37 to 65] | 59 [49 to 71] | 58 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 9 | 0 | 3 | 20
  Male | 3 | 4 | 2 | 5 | 7 | 6 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 4 | 6 | 16 | 6 | 6 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 7 | 4 | 6 | 15 | 6 | 6 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 4 | 6 | 16 | 6 | 6 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events Per Study Arm
Description: Safety and toxicity following vaccination with 7 long peptides in melanoma patients with and without TLR agonists.
  Patients are evaluated by safety labs and physical exams to assess for toxicity.
Time Frame: 6 months
Population: All participants enrolled and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1 + Part 2) | Arm F (Part 1) | Arm G(Part 1)
Number analyzed (Participants) | 5 | 7 | 4 | 6 | 16 | 6 | 6
Participants
  BLOOD/LYMPHATIC - Other | 0 | 0 | 0 | 0 | 1 | 0 | 0
  EAR/LABYRINTH - Tinnitus | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GASTROINTESTINAL - Constipation | 0 | 0 | 0 | 0 | 1 | 1 | 0
  GASTROINTESTINAL - Diarrhea | 1 | 1 | 0 | 0 | 0 | 2 | 1
  GASTROINTESTINAL - Mucositis oral | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GASTROINTESTINAL - Nausea | 1 | 0 | 1 | 2 | 5 | 2 | 2
  GASTROINTESTINAL - Other | 0 | 0 | 0 | 0 | 0 | 0 | 1
  GASTROINTESTINAL - Vomiting | 0 | 0 | 0 | 0 | 1 | 1 | 0
  GENERAL AND ADMINISTRATION SITE - Chills | 1 | 2 | 0 | 3 | 12 | 3 | 3
  GENERAL AND ADMINISTRATION SITE - Fatigue | 4 | 5 | 0 | 3 | 12 | 3 | 4
  GENERAL AND ADMINISTRATION SITE - Fever | 0 | 1 | 0 | 2 | 8 | 2 | 2
  GENERAL AND ADMINISTRATION SITE - Flu like symptoms | 0 | 1 | 0 | 3 | 1 | 1 | 2
  GENERAL AND ADMINISTRATION SITE - Injection site reaction | 5 | 6 | 1 | 6 | 15 | 6 | 6
  GENERAL AND ADMINISTRATION SITE - Localized edema | 0 | 0 | 0 | 0 | 1 | 0 | 1
  GENERAL AND ADMINISTRATION SITE - Other | 1 | 2 | 0 | 0 | 6 | 3 | 1
  GENERAL AND ADMINISTRATION SITE - Pain | 0 | 0 | 0 | 1 | 1 | 1 | 2
  IMMUNE SYSTEM - Autoimmune disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0
  INJURY/POISONING/PROCEDURAL - Bruising | 0 | 0 | 0 | 0 | 1 | 0 | 0
  INVESTIGATIONS - Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  INVESTIGATIONS - Weight loss | 0 | 0 | 0 | 0 | 0 | 1 | 0
  INVESTIGATIONS - White blood cell decreased | 0 | 0 | 0 | 0 | 2 | 0 | 0
  METABOLISM/NUTRITION - Anorexia | 1 | 0 | 0 | 0 | 2 | 1 | 0
  MUSCULOSKELETAL/CONNECTIVE TISSUE - Arthralgia | 1 | 2 | 0 | 1 | 6 | 0 | 4
  MUSCULOSKELETAL/CONNECTIVE TISSUE - Generalized muscle weakness | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MUSCULOSKELETAL/CONNECTIVE TISSUE - Myalgia | 3 | 2 | 0 | 2 | 7 | 1 | 0
  MUSCULOSKELETAL/CONNECTIVE TISSUE - Pain in extremity | 1 | 1 | 0 | 1 | 1 | 0 | 0
  MUSCULOSKELETAL/CONNECTIVE TISSUE - Other | 0 | 0 | 0 | 0 | 1 | 0 | 0
  NERVOUS SYSTEM - Dizziness | 1 | 0 | 0 | 2 | 2 | 0 | 1
  NERVOUS SYSTEM - Dysgeusia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  NERVOUS SYSTEM - Headache | 2 | 2 | 0 | 3 | 6 | 1 | 1
  PSYCHIATRIC - Anxiety | 0 | 0 | 0 | 0 | 0 | 1 | 0
  RESPIRATORY/THORACIC/MEDIASTINAL - Allergic rhinitis | 1 | 1 | 0 | 0 | 2 | 1 | 0
  RESPIRATORY/THORACIC/MEDIASTINAL - Cough | 0 | 1 | 0 | 0 | 1 | 0 | 2
  RESPIRATORY/THORACIC/MEDIASTINAL - Dyspnea | 0 | 0 | 0 | 1 | 0 | 0 | 0
  RESPIRATORY/THORACIC/MEDIASTINAL - Sore throat | 0 | 1 | 0 | 0 | 1 | 1 | 2
  SKIN/SUBCUTANEOUS TISSUE - Hyperhidrosis | 0 | 1 | 0 | 0 | 7 | 1 | 1
  SKIN/SUBCUTANEOUS TISSUE - Pain of skin | 0 | 0 | 0 | 0 | 0 | 0 | 1
  SKIN/SUBCUTANEOUS TISSUE - Pruritus | 1 | 0 | 0 | 0 | 0 | 1 | 0
  SKIN/SUBCUTANEOUS TISSUE - Rash maculo-papular | 0 | 1 | 0 | 1 | 0 | 0 | 1
  SKIN/SUBCUTANEOUS TISSUE - Scalp pain | 1 | 0 | 0 | 0 | 0 | 0 | 0
  SKIN/SUBCUTANEOUS TISSUE - Skin hyperpigmentation | 0 | 0 | 0 | 0 | 2 | 0 | 0
  SKIN/SUBCUTANEOUS TISSUE - Skin hypopigmentation | 0 | 0 | 0 | 0 | 0 | 1 | 0
  SKIN/SUBCUTANEOUS TISSUE - Skin induration | 4 | 2 | 1 | 0 | 14 | 2 | 5
  SKIN/SUBCUTANEOUS TISSUE - Skin ulceration | 0 | 0 | 0 | 0 | 1 | 0 | 2
  VASCULAR - Flushing | 0 | 0 | 0 | 0 | 5 | 0 | 1
  VASCULAR - Hot flashes | 0 | 0 | 1 | 2 | 1 | 2 | 2
  VASCULAR - Other | 0 | 0 | 0 | 0 | 1 | 0 | 0
  DLTs | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: T Cell Response in Peripheral Blood Over Duration of Study Participation
Description: Levels of peptide-reactive CD8+ T cells in the peripheral blood: number of participants with T cell response to minimal epitope for CD8 T cells. This was assessed by direct (ex vivo) IFN-gamma ELIspot assay for reactivity to known minimal epitopes. To be considered positive, there had to be an increase compared to the maximum negative control target by at least 2-fold and by at least 20 IFN-gamma secreting cells per 100,000 CD8 T cells evaluated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm E (Part 1): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  IFA: 2 mL administered half intradermally and half subcutaneously
  Except that one patient, on Part 2, received all 6 vaccines in the same skin site, and did not have tetanus peptide in the vaccine.
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1) | Arm F (Part 1) | Arm G(Part 1)
Number analyzed (Participants) | 5 | 7 | 4 | 6 | 16 | 6 | 6
Participants | 2 | 1 | 0 | 0 | 4 | 1 | 1

3. Secondary Outcome: T Cell Response and Function in Peripheral Blood
Description: CD4+ T cell responses to peptides in the vaccine, and their function
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm E (Part 1 + 2): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  IFA: 2 mL administered half intradermally and half subcutaneously
  Except that one participant on Arm E was on Part 2, where all vaccines were administered at the same vaccine site, and the tetanus peptide was not included in the vaccines.
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1 + 2) | Arm F (Part 1) | Arm G(Part 1)
Number analyzed (Participants) | 5 | 7 | 4 | 6 | 16 | 6 | 6
Participants | 4 | 3 | 0 | 1 | 8 | 1 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Description: All adverse events (treatment-related or not), All serious adverse events (treatment-related or not), and All Cause Mortality on study
Groups:
- Arm E (Part 1 + 2): Peptide Vaccine (LPV7) + Tetanus peptide + IFA + PolyICLC vaccines administered in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on Days 1, 8, 15, 36, 57, and 78.
  Peptide Vaccine (LPV7) + Tetanus peptide: 1.5 mL administered half intradermally and half subcutaneously.
  PolyICLC: 1 mL administered half intradermally and half subcutaneously
  IFA: 2 mL administered half intradermally and half subcutaneously
  Except that one participant on Part 2 did not have tetanus peptide in the vaccine, and that participants vaccines were all administered at the same vaccine site.
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Arm D (Part 1) | Arm E (Part 1 + 2) | Arm F (Part 1) | Arm G(Part 1)
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/7 | 1/4 | 2/6 | 1/16 | 0/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/4 | 0/6 | 0/16 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 4/4 | 6/6 | 16/16 | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Part 1) (N=5) | Arm B (Part 1) (N=7) | Arm C (Part 1) (N=4) | Arm D (Part 1) (N=6) | Arm E (Part 1 + 2) (N=16) | Arm F (Part 1) (N=6) | Arm G(Part 1) (N=6)
Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 2 | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 6 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 3 | 0 | 3 | 12 | 4 | 3
Fatigue (General disorders) | 4 | 5 | 0 | 3 | 12 | 3 | 4
Fever (General disorders) | 0 | 1 | 1 | 2 | 8 | 2 | 2
Flu-like symptoms (General disorders) | 0 | 1 | 0 | 3 | 1 | 1 | 2
Injection site reaction (General disorders) | 5 | 6 | 2 | 6 | 15 | 6 | 6
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 3 | 3 | 1 | 2
Other (General disorders) | 1 | 2 | 0 | 0 | 7 | 3 | 1
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1
weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
white blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 7 | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 3 | 7 | 2 | 0
Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 3 | 6 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Allergic rhinitis (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1 | 1 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 2 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 7 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Rash - maculopapular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1
scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 0 | 14 | 2 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 3 | 2 | 2 | 2
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Other (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Other (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Edema trunk (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Venous Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Other (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT02126579/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02126579/ICF_001.pdf